CLINICAL TRIAL: NCT02434471
Title: Single Breath Hold Abdominal MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00061735
Record Dates: First submitted 2015-04-28; First posted 2015-05-05 (Estimated); Results first posted 2018-05-31 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Abdominal MRI

ARMS (2):
- Breath hold Liver Acquisition with Volume Acquisition (LAVA) (No Intervention): Subjects will undergo abdominal MRI with LAVA with conventional breath holds (typically four or more breath holds) per standard of care.
- Respiratory-triggered T1w DISCO LAVA (Active Comparator): The study will acquire extra image sets using DISCO LAVA with one breath hold during the arterial imaging phase. No additional breath holds will be required.
  Interventions: Device: Respiratory-triggered T1w DISCO LAVA

INTERVENTIONS:
Device: Respiratory-triggered T1w DISCO LAVA — The study will acquire extra image sets using DISCO LAVA with one breath hold during the arterial imaging phase. No additional breath holds will be required.
  1. Respiratory-triggered T1w DISCO LAVA precontrast
  2. Respiratory-triggered T1w DISCO LAVA in the portal venous phase
  3. Respiratory-triggered T1w DISCO LAVA in the equilibrium phase
  Arms: Respiratory-triggered T1w DISCO LAVA

SUMMARY:
The purpose of this study is to evaluate a single breath hold abdominal MRI protocol and compare the image quality of respiratory triggered 3D T1-weighted images against conventional breath hold images.

ELIGIBILITY:
Inclusion Criteria:

* undergoing abdominal MRI

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa R Bashir, MD, Principal Investigator — Duke University
Locations (1):
- DukeUMC, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects did not continue participation in the study if their scans were cancelled or rescheduled outside of their hospitalization. Twenty enrolled subjects fell into this category.
Groups:
- Conventional Breath-held LAVA Then Respiratory Triggered Exams: All study subjects underwent an MRI exam including conventional breath-held LAVA imaging pre- and post-contrast, as well as respiratory-triggered DISCO imaging pre- and post-contrast
Period: Overall Study
Arm/Group | Conventional Breath-held LAVA Then Respiratory Triggered Exams
Started | 34
Completed | 25
Not Completed | 9
Not completed — Physician Decision | 9

BASELINE CHARACTERISTICS:
Population: Participants who completed the study
Groups:
- All Subjects: All study subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.94 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Motion Artifact Scores
Description: Three investigators will independently evaluate MRI examinations. They will assign motion scores between respiratory triggered and corresponding breath hold acquisitions. 1 = no motion artifact; 2 = minimal motion artifact, no effect on diagnostic quality; 3 = moderate motion artifact with some, but not severe, effect on diagnostic quality; 4 = severe motion artifact, images degraded but interpretable; and 5 = extensive motion artifact, images nondiagnostic.
Time Frame: During MRI, up to 60 minutes
Population: The same 25 subjects were used in both groups.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Respiratory-triggered T1w DISCO LAVA: The study will acquire extra image sets using DISCO LAVA with one breath hold during the arterial imaging phase. No additional breath holds will be required.
  Respiratory-triggered T1w DISCO LAVA: The study will acquire extra image sets using DISCO LAVA with one breath hold during the arterial imaging phase. No additional breath holds will be required.
  1. Respiratory-triggered T1w DISCO LAVA precontrast
  2. Respiratory-triggered T1w DISCO LAVA in the portal venous phase
  3. Respiratory-triggered T1w DISCO LAVA in the equilibrium phase
Arm/Group | Breath Hold Liver Acquisition With Volume Acquisition (LAVA) | Respiratory-triggered T1w DISCO LAVA
Number analyzed (Participants) | 25 | 25
scores on a scale | 1.8 (1.0) | 2.4 (0.9)
Statistical Analysis 1: Comparison: Breath Hold Liver Acquisition With Volume Acquisition (LAVA) vs Respiratory-triggered T1w DISCO LAVA; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.6

2. Primary Outcome: Noise Scores
Description: Three investigators will independently evaluate MRI examinations. They will assign noise scores between respiratory triggered and corresponding breath hold acquisitions. 1 = no noise artifact; 2 = minimal noise artifact, no effect on diagnostic quality; 3 = moderate noise artifact with some, but not severe, effect on diagnostic quality; 4 = severe noise artifact, images degraded but interpretable; and 5 = severe noise artifact, images nondiagnostic.
Time Frame: During MRI, up to 60 minutes
Population: The same 25 subjects were used for each group.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Breath Hold Liver Acquisition With Volume Acquisition (LAVA) | Respiratory-triggered T1w DISCO LAVA
Number analyzed (Participants) | 25 | 25
scores on a scale | 1.7 (0.6) | 1.8 (0.7)
Statistical Analysis 1: Comparison: Breath Hold Liver Acquisition With Volume Acquisition (LAVA) vs Respiratory-triggered T1w DISCO LAVA; Test type: Other; p = 0.83, Mixed Models Analysis; Mean Difference (Final Values) = 0.1

ADVERSE EVENTS:
Time Frame: 60 minutes
Groups:
- All Subjects: All subjects who completed the study
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT02434471/Prot_SAP_000.pdf